CLINICAL TRIAL: NCT00169351
Title: National Gilles De La Tourette Study Group
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: RBM0418
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Tourette syndrome is rare. In France, about 3000 patients have a severe form of the disease. The aim of this study is to collect clinical characteristics in 200 patients with Tourette syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome

Exclusion Criteria:

* severe cognitive disorders

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yves Agid, MD, PhD, Study Director — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-HÔPITAL PITIÉ-SALPETRIERE, Paris, France

REFERENCES:
- [Derived] Worbe Y, Mallet L, Golmard JL, Behar C, Durif F, Jalenques I, Damier P, Derkinderen P, Pollak P, Anheim M, Broussolle E, Xie J, Mesnage V, Mondon K, Viallet F, Jedynak P, Ben Djebara M, Schupbach M, Pelissolo A, Vidailhet M, Agid Y, Houeto JL, Hartmann A. Repetitive behaviours in patients with Gilles de la Tourette syndrome: tics, compulsions, or both? PLoS One. 2010 Sep 24;5(9):e12959. doi: 10.1371/journal.pone.0012959. PMID 20885982